CLINICAL TRIAL: NCT00771537
Title: HIV Testing & Womens Attitudes on HIV Vaccine Trials
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Gregory Zimet, Professor, Indiana University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 0601-09; R01NR010004 (NIH)
Record Dates: First submitted 2008-10-10; First posted 2008-10-13 (Estimated); Results first posted 2013-07-09 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2013-06

CONDITIONS: HIV
Keywords: HIV Testing; Persuasion; Health Communication; Clinical Trials Participation; Attitudes toward Health; Diagnostic Tests; Behavioral Research; Intervention Studies

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (16):
- Arm 1. Control PLUS Control (No Intervention)
- Arm 2. Control PLUS 1-Sided (Experimental): No message intervention control condition regarding HIV testing AND 1-Sided message intervention experimental condition regarding HIV vaccine clinical trial participation.
  Interventions: Behavioral: Message Sidedness
- Arm 3. Control PLUS 2-Sided Trivial (Experimental): No message intervention control condition regarding HIV testing AND 2-Sided trivial message experimental intervention condition regarding HIV vaccine clinical trial participation.
  Interventions: Behavioral: Message Sidedness
- Arm 4. Control PLUS 2-Sided Major (Experimental): No message intervention control condition regarding HIV testing AND 2-Sided Major message experimental intervention condition regarding HIV vaccine clinical trial participation.
  Interventions: Behavioral: Message Sidedness
- Arm 5. 1-Sided PLUS Control (Experimental): 1-Sided message intervention experimental condition regarding HIV testing AND No message intervention control condition regarding HIV vaccine clinical trial participation.
  Interventions: Behavioral: Message Sidedness
- Arm 6. 1-Sided PLUS 1-Sided (Experimental): 1-Sided message intervention experimental condition regarding HIV testing AND 1-Sided message intervention experimental condition regarding HIV vaccine clinical trial participation.
  Interventions: Behavioral: Message Sidedness
- Arm 7. 1-Sided PLUS 2-Sided Trivial (Experimental): 1-Sided message intervention experimental condition regarding HIV testing AND 2-Sided Trivial message intervention experimental condition regarding HIV vaccine clinical trial participation.
  Interventions: Behavioral: Message Sidedness
- Aim 8. 1-Sided PLUS 2-Sided Major (Experimental): 1-Sided message intervention experimental condition regarding HIV testing AND 2-Sided Major message intervention experimental condition regarding HIV vaccine clinical trial participation.
  Interventions: Behavioral: Message Sidedness
- Arm 9. 2-Sided Trivial PLUS Control (Experimental): 2-Sided Trivial message intervention experimental condition regarding HIV testing AND No message intervention control condition regarding HIV vaccine clinical trial participation.
  Interventions: Behavioral: Message Sidedness
- Arm 10. 2-Sided Trivial PLUS 1-Sided (Experimental): 2-Sided Trivial message intervention experimental condition regarding HIV testing AND 1-Sided message intervention experimental condition regarding HIV vaccine clinical trial participation.
  Interventions: Behavioral: Message Sidedness
- Arm 11. 2-Sided Trivial PLUS 2-Sided Trivial (Experimental): 2-Sided Trivial message intervention experimental condition regarding HIV testing AND 2-Sided trivial message intervention experimental condition regarding HIV vaccine clinical trial participation.
  Interventions: Behavioral: Message Sidedness
- Arm 12. 2-Sided Trivial PLUS 2-Sided Major (Experimental): 2-Sided Trivial message intervention experimental condition regarding HIV testing AND 2-Sided major message intervention experimental condition regarding HIV vaccine clinical trial participation.
  Interventions: Behavioral: Message Sidedness
- Arm 13. 2-Sided Major PLUS Control (Experimental): 2-Sided major message intervention experimental condition regarding HIV testing AND No message intervention control condition regarding HIV vaccine clinical trial participation.
  Interventions: Behavioral: Message Sidedness
- Arm 14. 2-Sided Major PLUS 1-Sided (Experimental): 2-Sided major message intervention experimental condition regarding HIV testing AND 1-Sided message intervention experimental condition regarding HIV vaccine clinical trial participation.
  Interventions: Behavioral: Message Sidedness
- Arm 15. 2-Sided Major PLUS 2-Sided Trivial (Experimental): 2-Sided major message intervention experimental condition regarding HIV testing AND 2-Sided trivial message intervention experimental condition regarding HIV vaccine clinical trial participation.
  Interventions: Behavioral: Message Sidedness
- Arm 16. 2-Sided Major PLUS 2-Sided Major (Experimental): 2-Sided major message intervention experimental condition regarding HIV testing AND 2-Sided major message intervention experimental condition regarding HIV vaccine clinical trial participation.
  Interventions: Behavioral: Message Sidedness

INTERVENTIONS:
Behavioral: Message Sidedness — There are 16 pairs of messages varying in sidedness. Arm 1 is a no message control condition regarding HIV testing + a no message control condition regarding trial participation. Arm 2 is control + a 1-sided message. Arm 3 is control + a trivial 2-sided message. Arm 4 is control + a major 2-sided message. Arm 5 is a 1-sided message + a control. Arm 6 is a 1-sided message + a 1-sided message. Arm 7 is a 1-sided message + a trivial 2-sided message. Arm 8 is a 1-sided message + a major2-sided message. Arm 9 is a trivial 2-sided message + a control. Arm 10 is a trivial 2-sided message + a 1-sided message. Arm 11 is a trivial 2-sided message + a trivial 2-sided message. Arm 12 is a trivial 2-sided message + a major 2-sided message. Arm 13 is a major 2-sided message + a control. Arm 14 is a major 2-sided message + a 1-sided message. Arm 15 is a major 2-sided message + a trivial 2-sided message. Arm 16 is a major 2-sided message + a major2-sided message.
  Arms: Aim 8. 1-Sided PLUS 2-Sided Major; Arm 10. 2-Sided Trivial PLUS 1-Sided; Arm 11. 2-Sided Trivial PLUS 2-Sided Trivial; Arm 12. 2-Sided Trivial PLUS 2-Sided Major; Arm 13. 2-Sided Major PLUS Control; Arm 14. 2-Sided Major PLUS 1-Sided; Arm 15. 2-Sided Major PLUS 2-Sided Trivial; Arm 16. 2-Sided Major PLUS 2-Sided Major; Arm 2. Control PLUS 1-Sided; Arm 3. Control PLUS 2-Sided Trivial; Arm 4. Control PLUS 2-Sided Major; Arm 5. 1-Sided PLUS Control; Arm 6. 1-Sided PLUS 1-Sided; Arm 7. 1-Sided PLUS 2-Sided Trivial; Arm 9. 2-Sided Trivial PLUS Control

SUMMARY:
The purpose of this study is to test the effects of different persuasive informational messages on rates of rapid HIV testing and willingness to participate in a HIV vaccine clinical trial. Adult African-American, non-Latina White, and Latina women will be recruited. Women will initially be randomized to 4 groups: 1. no message control; 2. 1-sided message that mentions benefits of HIV testing; 3. 2-sided message that acknowledges minor opposition to testing, then refutes the opposition; and 4. 2-sided message that acknowledge stronger opposition to testing, then refutes the opposition. Women will be offered HIV testing, then re-randomized to a similar set of 4 messages related to HIV vaccine trials. There will therefore be 16 groups in total (4 X 4).

DETAILED DESCRIPTION:
This 5-year proposal responds to PAS-03-168, "Enrolling Women and Minorities in HIV/AIDS Research Trials." This study seeks to evaluate persuasive message interventions to increase HIV testing rates and improve acceptability of participation in a phase 3 HIV vaccine clinical trial among African-American, Latina, and White women. We plan to evaluate 1-sided messages, which mention only the benefits of an action, versus 2-sided messages, which mention negative aspects of the action, followed by positive counterarguments. The Health Belief Model, Inoculation and Attribution Theories will guide the research. Participants will be women attending urban community health clinics in Indianapolis, IN. Specific Aim 1 is to identify obstacles to HIV testing and to participation in a HIV vaccine clinical trial. This aim will be accomplished in years 1 and 2 through individual semi-structured interviews. We will analyze data via thematic content analysis and will use interview findings to assist in the development of measures and interventions employed in the intervention phase (years 3-5). Specific Aim 2 is to evaluate the effects of 2-sided versus 1-sided persuasive messages on rates of acceptance of rapid HIV testing. Demographic, behavioral, and attitudinal measures will be administered via audio computer-assisted self-interview (A-CASI). Participants will be randomized to the intervention groups via A-CASI as well. The outcome will be acceptance/rejection of free rapid HIV testing. This Aim will be evaluated via binary logistic regression. Specific Aim 3 is to evaluate the effects of 2-sided versus 1-sided messages on willingness to participate in phase 3 clinical trials for a preventive HIV vaccine. Participants will complete this 2nd A-CASI survey and will again be randomized to intervention groups. The outcome will be a scale measuring acceptability of clinical trial participation. This Aim will be evaluated via one-way Analysis of Variance. This study is relevant to public health in that the results may help us to understand how to improve enrollment of women and minorities into preventive HIV vaccine clinical trials and how to encourage women and minorities to get tested for HIV.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18 years of age or older
* Able to understand English or Spanish
* Able to give informed consent

Exclusion Criteria:

* Not female
* Under 18 years of age
* Not able to understand English and Spanish
* Unable to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2031 (Actual)
Dates: Start 2006-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory D Zimet, PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Medical Group Clinics, Indianapolis, Indiana, United States

REFERENCES:
- [Result] Burrage JW, Zimet GD, Cox DS, Cox AD, Mays RM, Fife RS, Fife KH. The Centers for Disease Control and Prevention revised recommendations for HIV testing: reactions of women attending community health clinics. J Assoc Nurses AIDS Care. 2008 Jan-Feb;19(1):66-74. doi: 10.1016/j.jana.2007.11.003. PMID 18191770
- [Derived] Kasting ML, Cox AD, Cox D, Fife KH, Katz BP, Zimet GD. The effects of HIV testing advocacy messages on test acceptance: a randomized clinical trial. BMC Med. 2014 Nov 6;12:204. doi: 10.1186/s12916-014-0204-4. PMID 25374047

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Message intervention details are in the Brief Summary
Groups:
- HIV TEST MSG Control/ VACCINE TRIAL MSG Control: No message intervention control condition regarding HIV testing AND No message intervention control condition regarding HIV vaccine clinical trial participation.
- HIV TEST MSG Control/ VACCINE TRIAL MSG 1-Sided: No message intervention control condition regarding HIV testing AND 1-Sided message intervention experimental condition regarding HIV vaccine clinical trial participation.
- HIV TEST MSG Control/ VACCINE TRIAL MSG 2-Sided Trivial: No message intervention control condition regarding HIV testing AND 2-Sided trivial message intervention experimental condition regarding HIV vaccine clinical trial participation.
- HIV TEST MSG Control/ VACCINE TRIAL MSG 2-Sided Major: No message intervention control condition regarding HIV testing AND 2-Sided major message intervention experimental condition regarding HIV vaccine clinical trial participation.
- HIV TEST MSG 1-Sided/ VACCINE TRIAL MSG Control: 1-Sided message intervention experimental condition regarding HIV testing AND No message intervention control condition regarding HIV vaccine clinical trial participation.
- HIV TEST MSG 1-Sided/ VACCINE TRIAL MSG 1-Sided: 1-Sided message intervention experimental condition regarding HIV testing AND 1-Sided message intervention experimental condition regarding HIV vaccine clinical trial participation.
- HIV TEST MSG 1-Sided/ VACCINE TRIAL MSG 2-Sided Trivial: 1-Sided message intervention experimental condition regarding HIV testing AND 2-Sided trivial message intervention experimental condition regarding HIV vaccine clinical trial participation.
- HIV TEST MSG 1-Sided/ VACCINE TRIAL MSG 2-Sided Major: 1-Sided message intervention experimental condition regarding HIV testing AND 2-Sided major message intervention experimental condition regarding HIV vaccine clinical trial participation.
- HIV TEST MSG 2-Sided Trivial/ VACCINE TRIAL MSG Control: 2-Sided Trivial message intervention experimental condition regarding HIV testing AND No message intervention control condition regarding HIV vaccine clinical trial participation.
- HIV TEST MSG 2-Sided Trivial/ VACCINE TRIAL MSG 1-Sided: 2-Sided Trivial message intervention experimental condition regarding HIV testing AND 1-Sided message intervention experimental condition regarding HIV vaccine clinical trial participation.
- HIV TEST MSG 2-Sided Trivial/ VACCINE TRIAL MSG 2-Sided Trivia: 2-Sided Trivial message intervention experimental condition regarding HIV testing AND 2-Sided trivial message intervention experimental condition regarding HIV vaccine clinical trial participation.
- HIV TEST MSG 2-Sided Trivial/ VACCINE TRIAL MSG 2-Sided Major: 2-Sided Trivial message intervention experimental condition regarding HIV testing AND 2-Sided major message intervention experimental condition regarding HIV vaccine clinical trial participation.
- HIV TEST MSG 2-Sided Major/ VACCINE TRIAL MSG Control: 2-Sided major message intervention experimental condition regarding HIV testing AND No message intervention control condition regarding HIV vaccine clinical trial participation.
- HIV TEST MSG 2-Sided Major/ VACCINE TRIAL MSG 1-Sided: 2-Sided major message intervention experimental condition regarding HIV testing AND 1-Sided message intervention experimental condition regarding HIV vaccine clinical trial participation.
- HIV TEST MSG 2-Sided Major/ VACCINE TRIAL MSG 2-Sided Trivial: 2-Sided major message intervention experimental condition regarding HIV testing AND 2-Sided trivial message intervention experimental condition regarding HIV vaccine clinical trial participation.
- HIV TEST MSG 2-Sided Major/ VACCINE TRIAL MSG 2-Sided Major: 2-Sided major message intervention experimental condition regarding HIV testing AND 2-Sided major message intervention experimental condition regarding HIV vaccine clinical trial participation.
Period: Overall Study
Arm/Group | HIV TEST MSG Control/ VACCINE TRIAL MSG Control | HIV TEST MSG Control/ VACCINE TRIAL MSG 1-Sided | HIV TEST MSG Control/ VACCINE TRIAL MSG 2-Sided Trivial | HIV TEST MSG Control/ VACCINE TRIAL MSG 2-Sided Major | HIV TEST MSG 1-Sided/ VACCINE TRIAL MSG Control | HIV TEST MSG 1-Sided/ VACCINE TRIAL MSG 1-Sided | HIV TEST MSG 1-Sided/ VACCINE TRIAL MSG 2-Sided Trivial | HIV TEST MSG 1-Sided/ VACCINE TRIAL MSG 2-Sided Major | HIV TEST MSG 2-Sided Trivial/ VACCINE TRIAL MSG Control | HIV TEST MSG 2-Sided Trivial/ VACCINE TRIAL MSG 1-Sided | HIV TEST MSG 2-Sided Trivial/ VACCINE TRIAL MSG 2-Sided Trivia | HIV TEST MSG 2-Sided Trivial/ VACCINE TRIAL MSG 2-Sided Major | HIV TEST MSG 2-Sided Major/ VACCINE TRIAL MSG Control | HIV TEST MSG 2-Sided Major/ VACCINE TRIAL MSG 1-Sided | HIV TEST MSG 2-Sided Major/ VACCINE TRIAL MSG 2-Sided Trivial | HIV TEST MSG 2-Sided Major/ VACCINE TRIAL MSG 2-Sided Major
Started | 135 | 124 | 151 | 114 | 127 | 118 | 128 | 132 | 115 | 119 | 133 | 137 | 128 | 124 | 124 | 122
Completed | 135 | 124 | 151 | 114 | 127 | 118 | 128 | 132 | 115 | 119 | 133 | 137 | 128 | 124 | 124 | 122
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- HIV TEST MSG Control/ VACCINE TRIAL MSG 2-Sided Trivial: No message intervention control condition regarding HIV testing AND 2-Sided trivial message experimental intervention condition regarding HIV vaccine clinical trial participation.
- HIV TEST MSG Control/ VACCINE TRIAL MSG 2-Sided Major: No message intervention control condition regarding HIV testing AND 2-Sided Major message experimental intervention condition regarding HIV vaccine clinical trial participation.
- Total: Total of all reporting groups
Arm/Group | HIV TEST MSG Control/ VACCINE TRIAL MSG Control | HIV TEST MSG Control/ VACCINE TRIAL MSG 1-Sided | HIV TEST MSG Control/ VACCINE TRIAL MSG 2-Sided Trivial | HIV TEST MSG Control/ VACCINE TRIAL MSG 2-Sided Major | HIV TEST MSG 1-Sided/ VACCINE TRIAL MSG Control | HIV TEST MSG 1-Sided/ VACCINE TRIAL MSG 1-Sided | HIV TEST MSG 1-Sided/ VACCINE TRIAL MSG 2-Sided Trivial | HIV TEST MSG 1-Sided/ VACCINE TRIAL MSG 2-Sided Major | HIV TEST MSG 2-Sided Trivial/ VACCINE TRIAL MSG Control | HIV TEST MSG 2-Sided Trivial/ VACCINE TRIAL MSG 1-Sided | HIV TEST MSG 2-Sided Trivial/ VACCINE TRIAL MSG 2-Sided Trivia | HIV TEST MSG 2-Sided Trivial/ VACCINE TRIAL MSG 2-Sided Major | HIV TEST MSG 2-Sided Major/ VACCINE TRIAL MSG Control | HIV TEST MSG 2-Sided Major/ VACCINE TRIAL MSG 1-Sided | HIV TEST MSG 2-Sided Major/ VACCINE TRIAL MSG 2-Sided Trivial | HIV TEST MSG 2-Sided Major/ VACCINE TRIAL MSG 2-Sided Major | Total
Number analyzed (Participants) | 135 | 124 | 151 | 114 | 127 | 118 | 128 | 132 | 115 | 119 | 133 | 137 | 128 | 124 | 124 | 122 | 2031
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 10
  Between 18 and 65 years | 126 | 115 | 137 | 104 | 119 | 111 | 121 | 124 | 111 | 112 | 126 | 128 | 118 | 120 | 118 | 119 | 1909
  >=65 years | 9 | 8 | 14 | 10 | 7 | 6 | 6 | 6 | 3 | 7 | 6 | 7 | 10 | 4 | 6 | 3 | 112
Age Continuous [Mean (Standard Deviation); unit: years] | 42 (14) | 44 (14) | 47 (13) | 45 (15) | 44 (13) | 44 (12) | 44 (14) | 45 (14) | 42 (13) | 44 (13) | 44 (13) | 43 (13) | 46 (13) | 44 (13) | 44 (12) | 42 (13) | 44 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 124 | 151 | 114 | 127 | 118 | 128 | 132 | 115 | 119 | 133 | 137 | 128 | 124 | 124 | 122 | 2031
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 135 | 124 | 151 | 114 | 127 | 118 | 128 | 132 | 115 | 119 | 133 | 137 | 128 | 124 | 124 | 122 | 2031

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Accepted Rapid HIV Testing.
Description: Acceptance of rapid HIV testing. Acceptance was assessed by actual administration of rapid oral HIV test by research staff.
Time Frame: During study visit. At approximately 30 minutes into the study visit. After part 1 of the questionnaire was completed.
Measure: Number; unit: participants
Groups:
- Control: No message intervention control condition regarding HIV testing AND No message intervention control condition regarding HIV vaccine clinical trial participation.
- 1-Sided: 1-Sided message intervention experimental condition regarding HIV testing AND No message intervention control condition regarding HIV vaccine clinical trial participation.
- 2-Sided Trivial: 2-Sided Trivial message intervention experimental condition regarding HIV testing AND No message intervention control condition regarding HIV vaccine clinical trial participation.
- 2-Sided Major: 2-Sided major message intervention experimental condition regarding HIV testing AND No message intervention control condition regarding HIV vaccine clinical trial participation.
Arm/Group | Control | 1-Sided | 2-Sided Trivial | 2-Sided Major
Number analyzed (Participants) | 524 | 505 | 504 | 498
participants | 458 | 401 | 410 | 418
Statistical Analysis 1: Comparison: Control vs 1-Sided; Test type: Superiority or Other; p = 0.05, Regression, Logistic; Odds Ratio (OR) = .69, 95% CI 2-sided [.50 to .96], Standard Error of Mean .17 — Women in the 1-sided message group accepted testing at a lower rate (79.4%) than those in the control group (87.4%)
Statistical Analysis 2: Comparison: Control vs 2-Sided Trivial; Test type: Superiority or Other; p = .10, Regression, Logistic; Odds Ratio (OR) = .75, 95% CI 2-sided [.54 to 1.04], Standard Error of Mean .17 — Women in the 2-sided trivial group were no different in their acceptance rate of HIV testing (81.3%) than women in the control group (87.4%)
Statistical Analysis 3: Comparison: Control vs 2-Sided Major; Test type: Superiority or Other; p = .63, Regression, Logistic; Odds Ratio (OR) = .92, 95% CI 2-sided [.65 to 1.30], Standard Error of Mean .176 — Women in the 2-sided major group were no different in rates of accepting HIV testing (83.9%) than women in the control group (87.4%)

2. Primary Outcome: Willingness to Participate in a HIV Vaccine Clinical Trial
Description: Willingness to Participate in a HIV Vaccine Clinical Trial. Assessed via participant self-report with 6 items on Part 2 of the questionnaire. Item responses measured on 5-point Likert-type scale ranging from Strongly Disagree (value = 1) to Strongly Agree (value = 5).
Time Frame: Approximately 60 minutes into the study visit, at the end of Part 2 of the questionnaire.
Population: Only participants who answered the Willingness to Participate questions on the survey were included in these analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Control/Control: No message intervention control condition regarding HIV testing AND No message intervention control condition regarding HIV vaccine clinical trial participation.
- 1-Sided: No message intervention control condition regarding HIV testing AND 1-Sided message intervention experimental condition regarding HIV vaccine clinical trial participation.
- 2-Sided Trivial: No message intervention control condition regarding HIV testing AND 2-Sided trivial message experimental intervention condition regarding HIV vaccine clinical trial participation.
- 2-Sided Major: No message intervention control condition regarding HIV testing AND 2-Sided Major message experimental intervention condition regarding HIV vaccine clinical trial participation.
Arm/Group | Control/Control | 1-Sided | 2-Sided Trivial | 2-Sided Major
Number analyzed (Participants) | 500 | 480 | 530 | 502
units on a scale | 2.46 (1.15) | 2.52 (1.18) | 2.55 (1.18) | 2.47 (1.12)
Statistical Analysis 1: Comparison: Control/Control vs 1-Sided; One-way Analysis of Variance; Test type: Superiority or Other; p < .60, ANOVA; Degrees of freedom = (1,978); Marginal Means = 2.49, 95% CI 2-sided [2.42 to 2.56], Standard Error of Mean .037 — There was no significant effect for the 1-sided message compared to the control group on Willingness to Participate in an HIV vaccine clinical trial
Statistical Analysis 2: Comparison: Control/Control vs 2-Sided Trivial; One-Way Analysis of Variance; Test type: Superiority or Other; p < .25, ANOVA; degrees of freedom = (1,1028); Marginal Means = 2.51, 95% CI 2-sided [2.44 to 2.58], Standard Error of Mean .036 — There was no significant effect for the 2-sided trivial message compared to the control group on Willingness to Participate in an HIV vaccine clinical trial
Statistical Analysis 3: Comparison: Control/Control vs 2-Sided Major; One-Way Analysis of Variance; Test type: Superiority or Other; p < .91, ANOVA; Marginal Means = 2.47, 95% CI 2-sided [2.40 to 2.54], Standard Error of Mean .036 — There was no significant effect for the 2-sided major message compared to the control group on Willingness to Participate in an HIV vaccine clinical trial

ADVERSE EVENTS:
Description: Adverse events were not collected.
Arm/Group | HIV TEST MSG Control/ VACCINE TRIAL MSG Control | HIV TEST MSG Control/ VACCINE TRIAL MSG 1-Sided | HIV TEST MSG Control/ VACCINE TRIAL MSG 2-Sided Trivial | HIV TEST MSG Control/ VACCINE TRIAL MSG 2-Sided Major | HIV TEST MSG 1-Sided/ VACCINE TRIAL MSG Control | HIV TEST MSG 1-Sided/ VACCINE TRIAL MSG 1-Sided | HIV TEST MSG 1-Sided/ VACCINE TRIAL MSG 2-Sided Trivial | HIV TEST MSG 1-Sided/ VACCINE TRIAL MSG 2-Sided Major | HIV TEST MSG 2-Sided Trivial/ VACCINE TRIAL MSG Control | HIV TEST MSG 2-Sided Trivial/ VACCINE TRIAL MSG 1-Sided | HIV TEST MSG 2-Sided Trivial/ VACCINE TRIAL MSG 2-Sided Trivia | HIV TEST MSG 2-Sided Trivial/ VACCINE TRIAL MSG 2-Sided Major | HIV TEST MSG 2-Sided Major/ VACCINE TRIAL MSG Control | HIV TEST MSG 2-Sided Major/ VACCINE TRIAL MSG 1-Sided | HIV TEST MSG 2-Sided Major/ VACCINE TRIAL MSG 2-Sided Trivial | HIV TEST MSG 2-Sided Major/ VACCINE TRIAL MSG 2-Sided Major
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No